CLINICAL TRIAL: NCT01369667
Title: Vitamin D and Immunomodulation: Effects in Crohn's Disease
Brief Title: Vitamin D Supplementation in Adult Crohn's Disease
Acronym: VITD-CD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Tara Raftery, Research dietitian, University of Dublin, Trinity College
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VITD/CD/01
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2011-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- vitamin D (Active Comparator): Capsule, one taken daily
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Capsule, one taken daily
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3
  Arms: vitamin D
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether vitamin D supplementation is effective in the prevention of relapse in Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients must fulfill the clinical criteria for diagnosis of Crohn's disease.
* Subjects must have inactive CD as defined by CDAI < 150
* CRP </=10 mg/L.

Exclusion Criteria:

* Pregnant and lactating women.
* Known hypersensitivity to vitamin D.
* Hypercalcaemia
* Current supplemental intake of vitamin D3 >800 IU/D.
* Diagnosis of any of the following: active tuberculosis, sarcoidosis, hyperparathyroidism, pseudohyperparathyroidism, renal failure or malignancy, active TB, sarcoidosis, lymphoma.
* Participation in a concurrent clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Clinical Relapse: defined as a CDAI of 150 or more and an increase in CDAI of more than 70 compared with baseline during the 12 month follow-up period. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Maria O'Sullivan, PhD, Principal Investigator — TCD
Locations (1):
- Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital,, Dublin, Ireland

REFERENCES:
- [Derived] O'Sullivan F, Raftery T, van Weele M, van Geffen J, McNamara D, O'Morain C, Mahmud N, Kelly D, Healy M, O'Sullivan M, Zgaga L. Sunshine is an Important Determinant of Vitamin D Status Even Among High-dose Supplement Users: Secondary Analysis of a Randomized Controlled Trial in Crohn's Disease Patients. Photochem Photobiol. 2019 Jul;95(4):1060-1067. doi: 10.1111/php.13086. Epub 2019 Mar 12. PMID 30649836